CLINICAL TRIAL: NCT06769386
Title: Investigation of Respiratory Muscle Strength, Respiratory Muscle Endurance and Muscle Oxygenation in Patients With Rheumatoid Arthritis
Brief Title: Investigation of Muscle Oxygenation in Patients With Rheumatoid Arthritis
Status: Recruiting | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Başak KAVALCI KOL, Principal Investigator, Kirsehir Ahi Evran Universitesi
Other Study IDs: AhiEvranU526
Record Dates: First submitted 2025-01-07; First posted 2025-01-10 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Rheumatoid Arthritis
Keywords: exercise capacity; muscle oxygenation; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rheumatoid Arthritis Group: Rheumatoid arthritis patients who are followed up in the Rheumatology Outpatient Clinic of the Department of Physical Medicine and Rehabilitation (diagnosed according to American College of Rheumatology/European Alliance of Associations for Rheumatology ACR/EULAR 2022 diagnostic criteria), aged between 18-65 years, and have a Disease Activity Score (DAS) -28 score below 2.6 in disease remission will be included.
- Control Group: As a control group, healthy individuals between the ages of 18-65, who are similar to the patients in terms of age and gender, without any disease, will be included in the study. Healthy individuals in the control group will be selected from volunteer colleagues, school friends, family and residential areas of the researchers to participate in the study.

SUMMARY:
The aim of this study is to investigate respiratory muscle strength, respiratory muscle endurance, muscle oxygenation, upper extremity and lower extremity exercise capacity in rheumatoid arthritis patients compared with healthy individuals.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic progressive autoimmune disease of unknown etiology with symmetric erosive synovitis and multisystem involvement. The disease causes significant long-term morbidity, reduced functional capacity, and increased mortality rates. Patients with rheumatoid arthritis avoid physical activity due to pain and fatigue. Despite the advances in pharmacological treatments in recent years, functional losses due to rheumatic diseases the resulting deterioration in quality of life, and loss of work continue. Physical inactivity is known to have detrimental effects on the cardiovascular and pulmonary systems by reducing muscle strength and aerobic capacity. The physiological reasons underlying skeletal muscle oxygenation that may cause muscle dysfunction in rheumatoid arthritis have not been investigated. In these patients, decreased arterial oxygen may reduce exercise capacity and cause muscle deoxygenation.

In rheumatoid arthritis patients, decreases in respiratory muscle strength, lung volumes, oxygen consumption, and six minute walk test distance cause cardiopulmonary deconditioning. Decreased exercise capacity increases the risk of cardiovascular disease and causes mortality in patients with RA.

This study aimed to, the effects of respiratory muscle strength, respiratory muscle endurance, upper and lower extremity muscle oxygenation, and upper and lower extremity exercise capacity in patients with stable disease activity.

ELIGIBILITY:
Rheumatoid Arthritis Group

Inclusion Criteria:

* Patients diagnosed with rheumatoid arthritis,
* The ages of 18-65 years,
* Volunteer to participate in the study will be included in the study.

Exclusion Criteria:

* Serious cardiopulmonary, neurological, neuromuscular, orthopedic and other systemic diseases or other diseases affecting physical functions,
* Participated in a planned exercise program in the last three months,
* Cognitive impairment that will cause difficulty in understanding and following exercise test instructions,
* Contraindications to exercise testing or exercise training according to the American Sports Medicine Association will not be included in the study.

Control Group

Inclusion Criteria:

* The ages of 18-65 years,
* Volunteer to participate in the study will be included in the study.

Exclusion Criteria:

* Diagnosed chronic or systemic disease,
* Regular exercise (physical activity) 3 days a week, 150 minutes/week of moderate intensity
* Smoking 10 packs x years or more,
* Pneumonia or any acute infection,
* Healthy individuals with any psychiatric disorder will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients (diagnosed according to American College of Rheumatology/European Alliance of Associations for Rheumatology ACR/EULAR 2022 diagnostic criteria) aged between 18-65 years, with a Disease Activity Score (DAS)-28 score below 2.6 in disease remission and followed up at the Rheumatology Polyclinic of the Department of Physical Medicine and Rehabilitation at Kirsehir Ahi Evran University will be included in the study.
  As a control group, healthy individuals between the ages of 18-65, who are similar to the patients in terms of age and gender, without any disease, will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2026-01-25 (Estimated); Study Completion 2027-01-25 (Estimated)

PRIMARY OUTCOMES:
Evaluation of respiratory muscle strength | First day
  An electronic mouth pressure measuring device that complies with American Thoracic Society and European Respiratory Society criteria will be used to assess respiratory muscle strength.
Evaluation of respiratory muscle endurance | First day
  The incremental threshold workload test will be used to assess respiratory muscle endurance.The PowerBreathe Wellness® (HaB International Ltd. Southam, United Kingdom) inspiratory muscle training device will be used in the incremental threshold load test.
Evaluation of Deltoid and Quadriceps Femoris Muscle Oxygenation | First and second day
  Muscle oxygen level of quadriceps femoris and deltoid muscles will be measured using Moxy® monitor (Moxy, Fortiori Design LLC, Minnesota, USA) before, during and after the six-minute walk test and six-minute peg-board and ring test.
Evaluation of Deltoid and Quadriceps Femoris Muscle Total Hemoglobin Level | First and second day
  Total hemoglobin level of quadriceps femoris and deltoid muscles will be measured using Moxy® monitor (Moxy, Fortiori Design LLC, Minnesota, USA) before, during and after the six-minute walk test and six-minute peg-board and ring test.

SECONDARY OUTCOMES:
Evaluation of submaximal exercise capacity | First day and second day
  The six-minute walk test will be performed according to American Thoracic Society criteria to evaluate functional exercise capacity.
Evaluation of upper extremity capacity | First day and second day
  The six-minute peg board and ring test will be used to assess upper extremity exercise capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Başak KAVALCI KOL, PhD, Principal Investigator — Kirsehir Ahi Evran Universitesi; Merve FIRAT, PhD, Study Chair — Kirsehir Ahi Evran Universitesi; Figen TUNCAY, Prof. Dr., Study Chair — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kırşehir Ahi Evran University, Physical Therapy and Rehabilitation Center, Cardiopulmonary Unit, Kırşehir, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All data will be stored in a locked cabinet.

REFERENCES:
- [Background] Wickerson L, Mathur S, Brooks D, Bonetti LV, Singer LG, Granton J, Reid WD. Skeletal muscle oxygenation and regional blood volume during incremental limb loading in interstitial lung disease. ERJ Open Res. 2020 Jan 27;6(1):00083-2019. doi: 10.1183/23120541.00083-2019. eCollection 2020 Jan. PMID 32010722
- [Background] Cimen B, Deviren SD, Yorgancloglu ZR. Pulmonary function tests, aerobic capacity, respiratory muscle strength and endurance of patients with rheumatoid arthritis. Clin Rheumatol. 2001;20(3):168-73. doi: 10.1007/s100670170058. PMID 11434466